CLINICAL TRIAL: NCT07354776
Title: A Randomized Controlled Trial Evaluating the Effects of Isometric Neck Exercises and Postural Advice on Cervicogenic Headache Symptoms , Serum Cortisol, and Brain-Derived Neurotrophic Factor Levels in Adolescents With Smartphone Addiction
Brief Title: Effect of Isometric Neck Exercises on Cervicogenic Headache, Cortisol, and BDNF in Adolescents With Smartphone Addiction
Acronym: CGH SPA BDNF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: The Institute of Physical Medicine and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2025/013
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cervicogenic Headache; Sleep Disturbance; Stress
Keywords: Exercise Physiology; Stress; Sleep disturbance; Isometric exercises
MeSH Terms: conditions — Post-Traumatic Headache; Parasomnias

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either an intervention group (receiving isometric neck exercises plus posture advice) or a control group (receiving posture advice only). Both groups will be followed in parallel over a one-month intervention period to assess changes in headache symptoms, stress biomarkers, sleep quality, and functional outcomes.
Who Masked: Participant
Masking Description: The coin flip for randomization is done by a researcher after a participant meets eligibility criteria and gives consent, ensuring group assignment happens at randomization. This method, though not using a pre-determined concealed sequence, reduces bias by preventing prediction of group assignment before eligibility is confirmed. Participants will be masked to group allocation. They will not be informed whether they are receiving only posture advice or posture advice combined with isometric neck exercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants receive a one-month supervised and home-based isometric neck exercise program combined with posture advice.
  Interventions: Behavioral: Isometric Neck Exercise Program
- Control Arm (Active Comparator): Participants receive posture advice only, with no exercise intervention.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Isometric Neck Exercise Program — One-month program of supervised (2x/week, 30 mins) and home-based (daily, 15 mins) exercises. Includes TENS, chin tucks, isometric neck exercises in multiple directions, head protrusion, wall push-ups, shoulder shrugs, weight-bearing shoulder flexion, and PNF for deep neck flexors. Combined with structured patient education on posture and smartphone ergonomics. Adherence supported via app reminders and weekly check-ins.
  Arms: Intervention Arm
Behavioral: Usual Care — Receives only basic posture advice with no structured exercises or ergonomic training.
  Arms: Control Arm

SUMMARY:
Cervicogenic headache (CGH) is a secondary headache type caused due to refereed pain arising from the cervical spine in the forehead, sometimes in temporal region. (1)Which may have great impact on our daily life activities; decreased range of motion at cervical spine, decreased sleep quality, increased stress, disturbed mood and altered physiologic chemicals. (2)It is found to be more prevalent in females and is experimentally diagnosed by the Cervical Flexion-Rotation Test (CFRT) which is performed by a therapist.(3) Also, the upper trapezius midpoint (2 cm lateral to C2) mostly acts as a pressure point.(4) Other pressure points in cervical region may also develop. The pain is mostly on one side and remains on one side. It can be dull aching or pressure like pain. No photophobia, phonophobia, nausea, or tearing of eyes is associated with it. (1)(5) In the modern age, smartphone addiction (SPA) contributes significantly to CGH by promoting forward head posture, rounded shoulders, and impaired proprioception. (4)Despite this, there is a clear gap in the literature regarding body awareness, ergonomics, and targeted prevention strategies for smartphone-related postural problems. There is an urgent need for structured training programs and therapeutic interventions to address these concerns, combined with long-term follow-up studies.(4) In this study, we focus on brain-derived neurotrophic factor (BDNF) as a key biomarker of pain sensitization. Chronic stress and pain, reduces neuronal BDNF uptake, decreasing the serum BDNF levels, (6)while effective interventions are expected to elevate BDNF levels, improving motor performance and reducing nociceptive signaling. (6)(7)Literature shows that there is a significant increase in BDNF levels in moderate intensity aerobic exercises groups as compared to control group.(7) We aim to improve BDNF levels through isometric targeted exercise and ultimately improving the synaptic plasticity, mitochondrial activity, increased beta-endorphins. Increase in body temperature through exercise will also reduce pain sensitization and improve function.

In this study we also target stress level by focusing on cortisol as a biomarker. As the physiological and psychological stress is increased due to prolong flexion and increased screen time sleep quality is also disturbed.(8) We aim to evaluate whether targeted isometric neck exercises can enhance BDNF levels, regulate cortisol as a stress marker, and ultimately improve CGH symptoms. As we know that high stress elevates cortisol and disrupts the HPA axis, (9)we hypothesize that exercise-induced adaptations will downregulate the HPA axis, decrease cortisol, restore neuronal health, and enhance cognitive and motor functions and we also address how poor sleep, exacerbated by excessive screen time, contributes to cognitive, memory, and metabolic issues. By investigating the effects of exercise on sleep quality, our study fills a crucial research gap linking SPA, stress, BDNF, cortisol, and CGH offering a novel therapeutic approach that combines patient education, circadian rhythm alignment, and structured isometric exercise to improve health outcomes in adolescents.

DETAILED DESCRIPTION:
Smartphone addiction (SPA) increasingly contributes to cervicogenic headaches (CGH) and alters stress biomarkers (cortisol, BDNF) in adolescents. We aim to evaluate isometric neck exercises' impact on CGH symptoms, cortisol, and BDNF levels in SPA-affected adolescents. It will be a single-blind randomized controlled trial (RCT). We calculated our sample size based on medium effect size as 0.9 with 80% power to be 44. Which include adolescents (13 to 24 years) with SPA and CGH.

Intervention: One month of supervised/home-based isometric neck exercises (n=24) versus control (n=24).

Outcomes: Primary: Changes in NDI, HIT-6. Secondary: Changes in cortisol, BDNF, PSQI from baseline to 1-month.

This RCT will assess if isometric exercises reduce CGH symptoms and modulate key biomarkers such as BDNF informing interventions for SPA-related health issues.

The primary outcome for this study was the reduction in Cervicogenic Headache (CGH) symptom burden and associated pain sensitization processes involved in causing CGH. This outcome will be quantified by measuring the change from baseline to 1-month post-intervention using three distinct measures:

* The Neck Disability Index (NDI): A questionnaire assessing perceived functional disability related to neck issues.
* The Headache Impact Test (HIT-6): A questionnaire evaluating the impact of headaches on daily function.
* Serum Brain-Derived Neurotrophic Factor (BDNF) levels: Determined via ELISA analysis, utilized as a biomarker potentially reflecting changes in neuronal plasticity associated with pain sensitization.

The secondary outcome will be stress reduction, evaluated via both physiological and subjective indicators linked to stress levels. This will be quantified by measuring the change from baseline to 1-month post-intervention using:

* Serum Cortisol levels: Determined via ELISA analysis, serving as a physiological marker of hypothalamic-pituitary-adrenal (HPA) axis activity.
* The Pittsburgh Sleep Quality Index (PSQI): A questionnaire assessing subjective sleep quality, considered here as an indicator influenced by overall stress. The Intervention Group (n=22) will participate in supervised exercise sessions twice weekly at the IPMR KMU Physiotherapy Department, each lasting 30 minutes and led by a physiotherapist. These sessions will include specific exercises:

TENS (for pain relief): Intensity is typically set to a sensory level, where the patient feels a comfortable tingling or buzzing sensation without muscle contraction. Pulse duration often ranges from 50-100 microseconds, and treatment sessions usually last for 20-30 minutes, performed once or twice daily.

Chin tuck in Gently retract chin backward ("double chin") while sitting or standing tall, keeping eyes forward. Low intensity, focusing on controlled muscle activation. Aims to strengthen deep neck muscles, improve posture, and stretch sub occipital muscles. Repetitions 10 times and hold times 10 sec and then released.

Isometric exercises involve contracting neck muscles against a fixed resistance (like your hand or a wall) in various directions (flexion, extension, lateral flexion, rotation) for 10-second holds. Performed at a moderate intensity for 10 repetitions, lasting about 15 minutes, this strengthening exercise aims to build neck muscle strength and endurance.

Head protrusion in antigravity Lying down with head slightly off the edge, actively lift head to neutral or hold isometrically against gravity for 10 seconds, repeated 5 times at moderate intensity. This exercise strengthens deep neck flexors and improves postural endurance.

Wall Push-Ups Standing facing a wall with hands shoulder-width apart, lean in by bending elbows, then push back. Intensity is moderate. Aims to strengthen chest, triceps, and key scapular stabilizers (serratus anterior, rhomboids, trapezius) for better shoulder posture. Reps 10 times Isometric shoulder shrugs by Standing or sitting tall, the individual actively elevates (shrugs) their shoulders straight up towards their ears, then lowers them back down by holding a weight of intensity is mild to moderate hold for 10 sec and repeat 6-10 times Weight-Bearing Shoulder Flexion: In supine position with both hands holding a stick/ weight raise arm forward and upward for 10 repetitions at moderate intensity. This functional exercise strengthens shoulder flexion and improves scapular/core stability under load, promoting integrated movement. Deep neck flexors engage to stabilize the head and neck against the shifting weight and forces during the arm movement.

PNF exercise for deep neck flexors in sitting position tuck chin towards the chest until you feel a mild to moderate stretch at the back of your neck.

Therapist will apply resistance in this position to engage your deep neck flexors in isometric contraction against the slight resistance for 10 sec then completely relax your neck muscles. Repeat this isometric contraction and relaxation of deep flexors 6-10 times.

Participants will perform the same exercises daily at home for approximately 15 minutes.

Patient education on posture and smartphone ergonomics. Adherence will be supported through app reminders and weekly phone check-ins, aiming for over 80% compliance.

where as controlled group will only receive posture advice subjective sleep quality, considered here as an indicator influenced by overall stress.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 13 to 19 years.
* Smartphone addiction, defined as using a smartphone for ≥4 hours per day.
* A confirmed diagnosis of Cervicogenic Headache (CGH), as determined by a positive Cervical Flexion-Rotation Test (CFRT) performed by a physical therapist.

Exclusion Criteria:

* Diagnosis of other primary headache disorders (e.g., migraine, tension-type headache, cluster headache) or sinusitis.
* Presence of fever, cranial tumors, meningitis, or subarachnoid hemorrhage.
* Known carotid or vertebral artery dysfunction.
* Significant use of other screened devices (e.g., tablets, laptops) that would confound the primary exposure.
* History of prior neck injuries or cervical fractures.
* Any medical condition that renders the individual unfit to participate in a moderate exercise program.
* Presence of photophobia or phonophobia.
* Current drug addiction.
* Extreme, uncorrectable vision issues (Snellen chart score worse than 20/200 in either eye).

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) Score | Change from Baseline to 1-month post-intervention
  The Neck Disability Index (NDI) is a 10-item questionnaire assessing perceived functional disability related to neck issues. The change in total score will be used to measure the impact of the intervention on neck-related function in adolescents with cervicogenic headache.
Change in Headache Impact Test (HIT-6) Score | Change from Baseline to 1-month post-intervention.
  The Headache Impact Test (HIT-6) is a 6-item questionnaire evaluating the impact of headaches on daily function and quality of life. The change in total score will be used to measure the reduction in headache burden.
Change in Serum Brain-Derived Neurotrophic Factor (BDNF) Level | Change from Baseline to 1-month post-intervention.
  Serum BDNF levels, determined via ELISA analysis, will be used as a biomarker potentially reflecting changes in neuronal plasticity associated with pain sensitization in cervicogenic headache.

SECONDARY OUTCOMES:
Change in Serum Cortisol Level | Change from Baseline to 1-month post-intervention.
  Serum cortisol levels, determined via ELISA analysis, will serve as a physiological marker of hypothalamic-pituitary-adrenal (HPA) axis activity to evaluate the intervention's effect on physiological stress.
Change in Pittsburgh Sleep Quality Index (PSQI) Score | Change from Baseline to 1-month post-intervention.
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire assessing subjective sleep quality over a one-month interval. The change in global score will be used as an indicator influenced by overall stress and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ali Syed, Principal Investigator — Khyber Medical University; Mohsin Shah, Principal Investigator — Khyber Medical University Peshawar, Pakistan
Locations (1):
- Institute of Basic Medical Sciences (IBMS), Khyber Medical University, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in the primary publication (thesis and any subsequent journal articles) may be shared with qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available starting 6 months after the publication of the primary thesis findings (expected circa mid-2026). Data will be available for a period of 5 years.
Access Criteria: Access to data will be granted to qualified researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Proposals should be directed to the corresponding author (Dr. Mohsin Shah, Mohsin.ibms@kmu.edu.pk). A signed data access agreement will be required. Requestors will bear any associated costs.

REFERENCES:
- [Background] Aabroo S, Shafique S, Javed A, Fatima A, Khan O, Riaz S. Frequency of Cervicogenic Headache in Students Due To Usage of Smart Devices - Cross Sectional Survey. Pakistan J Rehabil. 2022;11(2):36-41
- [Background] Hall T, Briffa K, Hopper D. Clinical evaluation of cervicogenic headache: a clinical perspective. J Man Manip Ther. 2008;16(2):73-80. doi: 10.1179/106698108790818422. PMID 19119390
- [Background] Li W, Liu Y, Deng J, Wang T. Influence of aerobic exercise on depression in young people: a meta-analysis. BMC Psychiatry. 2024 Aug 20;24(1):571. doi: 10.1186/s12888-024-06013-6. PMID 39164715
- [Background] Blandini F, Rinaldi L, Tassorelli C, Sances G, Motta M, Samuele A, Fancellu R, Nappi G, Leon A. Peripheral levels of BDNF and NGF in primary headaches. Cephalalgia. 2006 Feb;26(2):136-42. doi: 10.1111/j.1468-2982.2005.01006.x. PMID 16426267
- [Background] Sadeghi A, Rostami M, Ameri S, Karimi Moghaddam A, Karimi Moghaddam Z, Zeraatchi A. Effectiveness of isometric exercises on disability and pain of cervical spondylosis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Jun 16;14(1):108. doi: 10.1186/s13102-022-00500-7. PMID 35710510